CLINICAL TRIAL: NCT05719792
Title: Comparison of the Effectiveness of Erector Spina Plane Block and Transforaminal Anterior Epidural Steroid Injections in Lumbar Radicular Pain
Brief Title: Comparison of the Effectiveness of Erector Spina Plane Block and Transforaminal Anterior Epidural Injections
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MU-SK-YO-17.01.23
Record Dates: First submitted 2023-01-16; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Lumbar Disc Herniation; Radiculopathy Lumbar
Keywords: Lumbar Transforaminal Epidural Injection; Erector Spinae Plane Block
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Those who had lumbar radicular pain: Patients with lumbar radicular pain identified by inclusion and exclusion criteria
  Interventions: Procedure: Transforaminal Epidural Steroid Injection; Procedure: Erector Spina Plane Block

INTERVENTIONS:
Procedure: Transforaminal Epidural Steroid Injection — In the TFESI group, all patients were positioned prone. The injection site was cleaned with povidone-iodine 3 times and a sterile drape was applied. Short-acting local anesthesia (3 mL of 2% prilocaine) was applied to the skin and subcutaneous tissue. A 3.5-inch, 22-gauge spinal needle was inserted just below the pedicle. It was advanced into the subpedicular space using the coaxial technique under the intermittent guidance of fluoroscopy. The needle position was confirmed through a lateral view. Using lateral views, the needle was placed at the posterior one-third of the foramen. Using the anteroposterior view, one to 2 mL of the contrast agent (300 mg/50 mL iohexol) was given and the distribution pattern was visualized. Once the epidural distribution of the contrast agent was confirmed without vascular flow, a mixture of 8 mg (two mL) of dexamethasone, 2 mL of physiological saline, and 1 mL (0.5%) of bupivacaine hydrochloride was injected.
Procedure: Erector Spina Plane Block — Patients are placed in the prone position to determine the vertebrae in the middle of the involved area. Following the provision of aseptic conditions, the spinous process of the vertebral midline is visualized using a high-frequency (8 MHz) linear ultrasound (USG) probe. The transverse process is, then, visualized approximately at the 3 cm lateral from the midline and the erector spinae muscle is visualized on it. The 22-gauge 50 mm block needle is advanced towards the in-plane section craniocaudally and the transverse process is touched. Then the needle is then withdrawn minimally to confirm that it is between the erector spinae muscle and the transverse process through hydrodissection. Following that, 5 mL from 0.5% bupivacaine hydrochloride, 8 mg dexamethasone and 3 ml saline is administered and local anesthetic spread is confirmed by USG.

SUMMARY:
Low back pain is one of the leading causes of disability and its social burden and economic cost are quite high. The lifetime prevalence in the population is frequently reported between 40% and 70%. Although there are many reasons that can lead to low back pain, radicular pain, which develops mostly secondary to lumbar disc hernia, is one of the most common pathologies.

Epidural corticosteroid and local anesthetic injections are an important treatment option in the treatment of lumbar radicular pain that does not respond to conservative methods. epidural injections; includes transforaminal, interlaminar and caudal approaches. The advantage of the transforaminal approach is that it allows access to the anterior epidural area, which is the region of pathology, and that it can spread to the target specifically around the inflamed nerve roots. The standard imaging technology used for steroid injections with this approach is fluoroscopy.

However, the aforementioned approaches carry the risk of dural puncture, epidural hematoma, epidural abscess, nerve damage, paralysis and many complications. In addition, radiation exposure is another problem. It may be possible to avoid a significant part of these risks by applying interfacial blocks used in regional anesthesia and postoperative pain control in the lumbar region. Recently, Erector Spina Plan Block (ESPB), an interfascial block technique, has been frequently applied under ultrasound (US) guidance as an alternative method to conventional paravertebral block. Investigators also frequently refer to this procedure in the clinic for patients with lumbar radicular pain.

In the literature, there are case reports of lumbar ESPB applied to patients with radicular pain due to disc herniation. Beyond case-level reports, there is no clinical study investigating the efficacy of this procedure technique for applications in the lumbar region. Starting from here, the aim of this study is; Investigators determined to compare the efficacy of erector spina plane block and transforaminal anterior epidural steroid injections in patients with radicular pain due to lumbar disc herniation.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Radicular low back pain
* Failure to respond to conservative treatments
* Single level lumbar nerve root compression due to disc herniation
* Agree to participate in the research

Exclusion Criteria:

* Patients younger than 18 years and older than 65 years
* Those with non-radicular low back pain
* Those with nerve root compression due to reasons other than disc herniation
* Those with Modic type-1 changes in lumbar MRI
* Those with spinal stenosis or spondylolisthesis
* Those diagnosed with spondylodiscitis
* Pregnant
* Those with inflammatory rheumatic disease
* Patients whose use of non-steroidal anti-inflammatory drugs is contraindicated (renal failure, bleeding disorders, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group will consist of patients who are planned to receive transforaminal epidural steroid injection or erector spina plane block treatment by the clinician, and who want to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in NRS (Numeric Rating Scale) | at first hour, at three weeks, at 3 months, at 6 months
  ≥50% reduction in the NRS scores at month 6 relative to the initial NRS scores.
Change in ODI (Oswestry Disability Index) | at first hour, at three weeks, at 3 months, at 6 months
  ≥40% reduction in ODI scores at month 6 relative to the initial ODI scores.
  (ODI is a deficiency/competence index that includes assessments grouped according to the types of daily activities in patients with low back pain.)

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghahreman A, Ferch R, Bogduk N. The efficacy of transforaminal injection of steroids for the treatment of lumbar radicular pain. Pain Med. 2010 Aug;11(8):1149-68. doi: 10.1111/j.1526-4637.2010.00908.x. PMID 20704666
- [Background] Manchikanti L, Benyamin RM, Falco FJ, Kaye AD, Hirsch JA. Do Epidural Injections Provide Short- and Long-term Relief for Lumbar Disc Herniation? A Systematic Review. Clin Orthop Relat Res. 2015 Jun;473(6):1940-56. doi: 10.1007/s11999-014-3490-4. PMID 24515404
- [Background] Celik M, Tulgar S, Ahiskalioglu A, Alper F. Is high volume lumbar erector spinae plane block an alternative to transforaminal epidural injection? Evaluation with MRI. Reg Anesth Pain Med. 2019 Apr 16:rapm-2019-100514. doi: 10.1136/rapm-2019-100514. Online ahead of print. No abstract available. PMID 30992410